CLINICAL TRIAL: NCT00234767
Title: Economic Analysis of Pulmonary Artery Catheter Use (EA-PAC)
Brief Title: Study of the Economics of Pulmonary Artery Catheter Use in Patients With Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: R01HS011620 (AHRQ)
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Lung Diseases
Keywords: Acute Respiratory Distress Syndrome; ARDS; Acute Lung Injury; ALI; Cost-effectiveness; Pharmacoeconomics; Long-term follow-up
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Lung Diseases

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Pulmonary Artery Catheter
Behavioral: Protocolized Fluid Management

SUMMARY:
Study of the long term outcomes and economic impact of the pulmonary artery catheter in acute respiratory distress syndrome (ARDS/ALI) patients.

DETAILED DESCRIPTION:
The pulmonary artery catheter (PAC) is a commonly used device that provides hemodynamic data to guide care of the critically ill, such as patients with acute lung injury or the acute respiratory distress syndrome (ARDS/ALI). Clinicians believe PAC use improves decision-making and patient outcomes but evidence is lacking and recent data suggest the PAC may increase mortality as well as considerably increasing costs. In response, the NHLBI funded a large multicenter trial (Fluid And Catheter Treatment Trial (FACTT) (N01-HR-46054-46064)) where ARDS/ALI patients were randomized to receive a PAC or the less invasive central venous catheter (CVC) and received a liberal or conservative fluid management protocol in response to data provided by the PAC or CVC. The primary end-point is in-patient mortality.

We are complementing FACTT with a concurrent economic analysis of the PAC. Our aims are to: 1.) compare differences between study arms in long-term survival, quality of life, and quality-adjusted survival; 2.) compare differences between study arms in acute care and long-term costs; 3.) calculate the cost-efficacy of PAC use (i.e., the balance of costs and effects under the controlled environment of the FACTT trial), and; 4.) estimate cost-effectiveness under more "real-world" conditions and produce life-time cost-effectiveness ratios, thereby facilitating comparison of our results to other cost-effectiveness analyses.

We are achieving Aims 1-3 by augmenting FACTT data collection with detailed information on hospital costs, extended survival follow-up for a minimum of one year, and post-discharge patient interviews to determine quality of life and resource use in the first year. We will achieve Aim 4 by constructing a microsimulation model first calibrated by results from FACTT and published data on life-expectancy and costs and then adjusted to reflect the broader patient case-mix and clinical effects of PAC use in routine clinical practice. We are using patient-level data from the King County Lung Injury Project epidemiology study (NHLBI HL-96-014) to adjust case-mix and patient-level data from a large pragmatic trial of PAC use in the United Kingdom to adjust the clinical effects of PAC use.

The results of our adjunct to FACTT will substantially amplify the value of the data being collected and provide, for the first time, robust estimates from randomized data of the economic effects of the widespread application of this important technology.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Fluid and Catheter Treatment Trial (FACTT)

Exclusion Criteria:

* Did not consent to economic substudy and long-term follow-up

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650
Dates: Start 2001-09; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek C Angus, MD, MPH, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Derived] Clermont G, Kong L, Weissfeld LA, Lave JR, Rubenfeld GD, Roberts MS, Connors AF Jr, Bernard GR, Thompson BT, Wheeler AP, Angus DC; NHLBI ARDS Clinical Trials Network. The effect of pulmonary artery catheter use on costs and long-term outcomes of acute lung injury. PLoS One. 2011;6(7):e22512. doi: 10.1371/journal.pone.0022512. Epub 2011 Jul 21. PMID 21811626
- See also: CRISMA Laboratory Webpage- CRISMA coordinates the EA-PAC study — http://www.ccm.upmc.edu/research/res_crisma.html